CLINICAL TRIAL: NCT07087977
Title: Holmium:YAG Laser With MOSES Technology vs Thulium Fiber Laser in Supine Mini-percutaneous Nephrolithotomy With Vacuum-assisted Renal Access Sheath: A Prospective, Randomized Clinical Trial
Brief Title: HoYAG vs TFL in miniPCNL With ClearPetra
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Bristol Whiles, MD, Assistant Professor of Urology, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00161413
Record Dates: First submitted 2025-05-30; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Nephrolithiasis; Kidney Stone
Keywords: Nephrolithiasis; Kidney Stone; ClearPetra; HoYAG; TFL
MeSH Terms: conditions — Nephrolithiasis; Kidney Calculi

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- MiniPCNL with HoYAG (Active Comparator): In Arm 1, participants will undergo miniPCNL with ClearPetra™ vacuum-assisted ureteral access sheath with HoYAG laser platform. Participants will undergo miniPCNL per standard of care
  Interventions: Device: HoYAG laser
- MiniPCNL with TFL (Active Comparator): In Arm 2, participants will undergo miniPCNL with ClearPetra™ vacuum-assisted ureteral access sheath with TFL laser platform. Participants will undergo miniPCNL per standard of care
  Interventions: Device: TFL laser platform

INTERVENTIONS:
Device: HoYAG laser — Patients will be randomly assigned (1:1) to HoYAG laser or TFL laser group for miniPCNL surgery according to standard of care.
  Arms: MiniPCNL with HoYAG
Device: TFL laser platform — Patients will be randomly assigned (1:1) to HoYAG or TFL laser group for MiniPCNL surgery according to standard of care.
  Arms: MiniPCNL with TFL

SUMMARY:
Mini percutaneous nephrolithotripsy is the treatment of choice for kidney stones over 2cm. This procedure commonly uses laser energy for breaking the stones, and among possible laser platforms, Hoyag and thulium fiber laser are FDA approved. Recently, this procedure has also included the use of vacuum assisted renal access sheaths, which allows suction to be employed together with the breaking of stones. This study intends to compare outcomes when using either laser platforms with suction sheaths in participants undergoing mini percutaneous nephrolithotripsy for the treatment of kidney stones.

DETAILED DESCRIPTION:
Due to the reduced diameter sheath of miniaturized percutaneous nephrolithotripsy (miniPCNL), surgical outcomes commonly rely on stone fragmentation provided by a laser energy source. Holmium:yttrium-aluminum-garnet laser (HoYAG) has long been considered the gold-standard for lithotripsy, but this position has been challenged by the introduction of the thulium fiber laser (TFL) since its approval for clinical use in 2017. In the same manner, the recently developed ClearPetra™(MicroTech Endoscopy®, China) vacuum-assisted renal access sheath (VA-RAS) is a novel technology that allows for concomitant irrigation and suction during the procedure.

No prior studies to date have exclusively investigated mini-PCNL outcomes with Ho:YAG and TFL when using VA-RAS. This study addresses the literature paucity regarding the outcomes when utilizing the high-power Ho:YAG with MOSES technology vs. TFL in mini-PCNL with VA-RAS. This study hypothesizes that the Ho:YAG may provide more efficient stone clearance, secondary to its superior ability to fragment stones when compared to the TLF laser, which primarily dusts despite the laser settings utilized.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females over 18 years of age
2. Patients with kidney stones, with stone burden larger than 15 mm.
3. Patients undergoing new percutaneous access with primary, supine, unilateral mini-PCNL.

   Exclusion Criteria:
4. Simultaneous use of more than 1 laser platform or other form of fragmentation (e.g., ultrasonic).
5. Patients undergoing simultaneous treatment of contralateral kidney stones during the same procedure.
6. Patients undergoing simultaneous treatment of ureteral stones during the same procedure.
7. Pregnant patients.
8. Presence of genitourinary anatomical abnormalities.
9. Uncorrected coagulopathy.
10. External urinary catheters.
11. Immunosuppressed patients.
12. Non-elective procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Stone Lithotripsy time between HoYAG and TFL | Procedure
  Time from scope insertion to scope removal

SECONDARY OUTCOMES:
Total operative time between HoYAG and TFL | Procedure
  Time from time-out to procedure finish
Stone Free Status between ClearPetra and traditional approach | 90 days
  Stone free is defined as no residual stones larger than 2mm in post operative CT scan
Laser Energy | Procedure
  Laser efficiency will be measured by evaluating the laser energy in kilojoules used during the procedure.
Laser Time | Procedure
  Laser efficiency will be measured by evaluating the time in minutes the laser was used during the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Whiles, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li P, Huang Z, Sun X, Yang T, Wang G, Jiang Y, Ke C, Li J. Comparison of Vacuum Suction Sheath and Non-Vacuum Suction Sheath in Minimally Invasive Percutaneous Nephrolithotomy: A Meta-Analysis. J Invest Surg. 2022 May;35(5):1145-1152. doi: 10.1080/08941939.2021.1995538. Epub 2021 Dec 13. PMID 34902273
- [Background] Liu Y, Zhu W, Zeng G. Percutaneous nephrolithotomy with suction: is this the future? Curr Opin Urol. 2021 Mar 1;31(2):95-101. doi: 10.1097/MOU.0000000000000854. PMID 33470685
- [Background] Traxer O, Keller EX. Thulium fiber laser: the new player for kidney stone treatment? A comparison with Holmium:YAG laser. World J Urol. 2020 Aug;38(8):1883-1894. doi: 10.1007/s00345-019-02654-5. Epub 2019 Feb 6. PMID 30729311